CLINICAL TRIAL: NCT03502707
Title: A Randomized, Double-blind, Placebo-controlled Phase 1/2a Study for Safety and Immunogenicity Evaluations for Regimen Selection of Ad26.RSV.preF and/or RSV preF Protein Combinations Followed by Expanded Safety Evaluation in Adults Aged 60 Years and Older
Brief Title: A Study to Evaluate the Safety and Immunogenicity for Regimen Selection of Ad26.RSV.preF and/or RSV preF Protein Combinations Followed by Expanded Safety Evaluation in Adults Aged 60 Years and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR108456; VAC18193RSV1004 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (21):
- Cohort (C)1 Group (G)1: Placebo for RSV preF Protein (Placebo Comparator): Participants will receive intramuscular injection of placebo on Day 1, Day 57 and at Month 12.
  Interventions: Biological: Placebo
- C1 G2: RSV preF Protein (Experimental): Participants will receive intramuscular injection of 50 microgram (mcg) RSV preF protein on Day 1, Day 57 and at Month 12.
  Interventions: Biological: RSV preF Protein 50 mcg
- C1 G3: Placebo for Ad26.RSV.preF/RSV preF or RSV preF Protein (Placebo Comparator): Participants will receive intramuscular injection of placebo on Day 1, Day 57 and at Month 12.
  Interventions: Biological: Placebo
- C1 G4: Mixture of Ad26.RSV.preF/RSV preF Protein (Experimental): Participants will receive intramuscular injection of a mixture of 5*10^10 viral particles (vp) of Ad26.RSV.preF/RSV preF 50 mcg protein on Day 1, Day 57 and at Month 12.
  Interventions: Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 50 mcg
- C1 G5: RSV preF Protein (Experimental): Participants will receive intramuscular injection of 150 mcg RSV preF protein on Day 1, Day 57 and at Month 12.
  Interventions: Biological: RSV preF Protein 150 mcg
- C1 G6: Mixture of Placebo for Ad26.RSV.preF/RSV preF Protein (Placebo Comparator): Participants will receive intramuscular injection of placebo on Day 1, Day 57 and at Month 12.
  Interventions: Biological: Placebo
- C1 G7: Mixture of Ad26.RSV.preF/RSV preF Protein (Experimental): Participants will receive intramuscular injection of a mixture of 5*10^10 vp of Ad26.RSV.preF plus 150 mcg RSV preF protein on Day 1, Day 57 and at Month 12.
  Interventions: Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 150 mcg
- C1 G8: Placebo for Ad26.RSV.preF/Placebo for RSV preF Protein (Placebo Comparator): Participants will receive intramuscular injection of placebo on Day 1 and at Month 12 and in only 1 arm on Day 57.
  Interventions: Biological: Placebo
- C1 G9: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Participants will receive intramuscular injection of a mixture of 1*10^11 vp of Ad26.RSV.preF plus 150 mcg RSV preF protein in 1 arm on Day 1 and 57 and at Month 12 and placebo in another arm on Day 1 and at Month 12.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 150 mcg
- C1 G10: Ad26.RSV.preF, RSV preF Protein and Placebo (Experimental): Participants will receive separate intramuscular injections of 1*10^11 vp of Ad26.RSV.preF in 1 Arm and 150 mcg RSV preF protein in another arm on Day 1 and at Month 12 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: RSV preF Protein 150 mcg; Biological: Ad26.RSV.preF 1*10^11 vp
- C2 G11: Ad26.RSV.preF and Placebo (Experimental): Participants will receive intramuscular injection of 1*10^11 vp of Ad26.RSV.preF in 1 arm and placebo in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: Ad26.RSV.preF 1*10^11 vp
- C2 G12: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Participants will receive intramuscular injection of a mixture of 5*10^10 vp Ad26.RSV.preF plus 50 mcg RSV preF protein in 1 arm and placebo in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 50 mcg
- C2 G13: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Participants will receive intramuscular injection of a mixture of 1*10^11 vp Ad26.RSV.preF plus 50 mcg RSV preF protein in 1 arm and placebo in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 50 mcg
- C2 G14: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Participants will receive intramuscular injection of a mixture of 1*10^11 vp Ad26.RSV.preF plus 150 mcg RSV preF protein in 1 arm and placebo in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 150 mcg
- C2 G15: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Participants will receive intramuscular injection of a mixture of 5*10^10 vp Ad26.RSV.preF plus 150 mcg RSV preF protein in 1 arm and placebo in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 150 mcg
- C2 G16: Ad26.RSV.preF, RSV preF Protein and Placebo (Experimental): Data from C1 G10 will be pooled with those of C2 G16. Participants will receive separate intramuscular injections of 1*10^11 vp of Ad26.RSV.preF in 1 Arm and 150 mcg RSV preF protein in another arm on Day 1 and placebo in 1 arm on Day 57.
  Interventions: Biological: Placebo; Biological: RSV preF Protein 150 mcg; Biological: Ad26.RSV.preF 1*10^11 vp
- C2 G17: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo (Experimental): Data from C1 G9 will be pooled with those of C2 G17. Participants will receive intramuscular injection of a mixture of 1*10^11 vp of Ad26.RSV.preF plus 150 mcg RSV preF protein in 1 arm on Day 1 and 57 and placebo in another arm on Day 1.
  Interventions: Biological: Placebo; Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 150 mcg
- C2 G18: Placebo for Ad26.RSV.preF/Placebo for RSV preF Protein (Placebo Comparator): Participants will receive intramuscular injection of placebo in separate arms on Day 1 and in only 1 arm on Day 57.
  Interventions: Biological: Placebo
- C3 G19: Selected Regimen (SR) (Experimental): If a one-dose regimen is selected, participants in this group will receive SR on Day 1 and a booster (the SR) at Month 12 and month 24. The participants who are randomized to two-dose regimen will receive SR on Day 1 and Day 57, and a booster (the selected regimen) at Month 12.
  Interventions: Biological: Selected Regimen
- C3 G20: SR + Placebo for SR (Experimental): If a one-dose regimen is selected, participants in this group will receive SR on Day 1 and Month 24, and a placebo at Month 12. The participants who are randomized to two-dose regimen will receive selected regimen on Day 1 and Day 57, and a placebo at Month 12.
  Interventions: Biological: Placebo; Biological: Selected Regimen
- C3 G21: Placebo for SR (Placebo Comparator): If a one-dose regimen is selected, participants in this group will receive placebo for SR on Day 1 and at Month 12 and Month 24. The participants who are randomized to two-dose regimen will receive placebo for SR on Day 1, Day 57, and Month 12.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Placebo for Ad26.RSV.preF, RSV preF protein, Ad26.RSV.preF/RSV preF protein mixture and selected regimen will be administered as sterile saline for intramuscular injection.
  Arms: C1 G10: Ad26.RSV.preF, RSV preF Protein and Placebo; C1 G3: Placebo for Ad26.RSV.preF/RSV preF or RSV preF Protein; C1 G6: Mixture of Placebo for Ad26.RSV.preF/RSV preF Protein; C1 G8: Placebo for Ad26.RSV.preF/Placebo for RSV preF Protein; C1 G9: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G11: Ad26.RSV.preF and Placebo; C2 G12: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G13: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G14: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G15: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G16: Ad26.RSV.preF, RSV preF Protein and Placebo; C2 G17: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G18: Placebo for Ad26.RSV.preF/Placebo for RSV preF Protein; C3 G20: SR + Placebo for SR; C3 G21: Placebo for SR; Cohort (C)1 Group (G)1: Placebo for RSV preF Protein
Biological: RSV preF Protein 50 mcg — RSV preF will be administered as a solution for intramuscular injection at a dose of 50 mcg.
  Other Names: JNJ-64213175
  Arms: C1 G2: RSV preF Protein
Biological: RSV preF Protein 150 mcg — RSV preF will be administered as a solution for intramuscular injection at a dose of 150 mcg.
  Other Names: JNJ-64213175
  Arms: C1 G10: Ad26.RSV.preF, RSV preF Protein and Placebo; C1 G5: RSV preF Protein; C2 G16: Ad26.RSV.preF, RSV preF Protein and Placebo
Biological: Ad26.RSV.preF 1*10^11 vp — Ad26.RSV.preF will be administered as a solution for intramuscular injection at a dose of 1*10^11 vp.
  Other Names: JNJ-64400141
  Arms: C1 G10: Ad26.RSV.preF, RSV preF Protein and Placebo; C2 G11: Ad26.RSV.preF and Placebo; C2 G16: Ad26.RSV.preF, RSV preF Protein and Placebo
Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 50 mcg — Mixture of Ad26.RSV.preF (5*10^10 vp) and RSV preF protein (50 mcg) will be administered as a solution for intramuscular injection.
  Arms: C1 G4: Mixture of Ad26.RSV.preF/RSV preF Protein; C2 G12: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo
Biological: Mixture of Ad26.RSV.preF 5*10^10 vp Plus RSV preF Protein 150 mcg — Mixture of Ad26.RSV.preF (5*10^10 vp) and RSV preF protein (150 mcg) will be administered as a solution for intramuscular injection.
  Arms: C1 G7: Mixture of Ad26.RSV.preF/RSV preF Protein; C2 G15: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo
Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 50 mcg — Mixture of Ad26.RSV.preF (1*10^11 vp) and RSV preF protein (50 mcg) will be administered as a solution for intramuscular injection.
  Arms: C2 G13: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo
Biological: Mixture of Ad26.RSV.preF 1*10^11 vp Plus RSV preF Protein 150 mcg — Mixture of Ad26.RSV.preF (1*10^11 vp) and RSV preF protein (150 mcg) will be administered as a solution for intramuscular injection.
  Arms: C1 G9: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G14: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo; C2 G17: Mixture of Ad26.RSV.preF/RSV preF Protein and Placebo
Biological: Selected Regimen — A regimen from Cohort 1 or Cohort 2 will be selected and administered as a solution for intramuscular injection at the selected dose.
  Arms: C3 G19: Selected Regimen (SR); C3 G20: SR + Placebo for SR

SUMMARY:
The purpose of this study for:

Cohort 1 and Cohort 2: to assess the safety and reactogenicity of the intramuscular one- and two-dose regimens, with a booster at Month 12 (Cohort 1) and to select a regimen for Cohort 3.

Cohort 2 and part of Cohort 1: to assess respiratory syncytial virus (RSV) neutralizing antibody levels of the regimens containing RSV pre-fusion (preF) protein compared to the one-dose adenovirus serotype 26 respiratory syncytial virus pre-fusion (Ad26.RSV.preF) regimen.

Cohort 3: to assess the safety and reactogenicity of the selected regimen and a booster at Month 12 and/or Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Before randomization, a woman must be postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause) and not intending to conceive by any methods
* In the investigator's clinical judgment, participant must be either in good or stable health. Participants may have underlying illnesses such as hypertension, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms and signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* For participants in Cohorts 1 and 2 only: Participant must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the laboratory screening tests are outside the central laboratory normal reference ranges and additionally within the limits of toxicity Grade 2 according to the United States (US) Food and Drug Administration (FDA) toxicity, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant and appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* From the time of each vaccination through 3 months after each vaccination, participant agrees not to donate blood
* Participant must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Per serology testing in Cohorts 1 and 2 and per medical history in Cohort 3: Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Per serology testing in Cohorts 1 and 2 and per medical history in Cohort 3: Participant has human immunodeficiency virus (HIV) type 1 or type 2 infection
* Participant has had major psychiatric illness and/or drug or alcohol abuse which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures
* Participant has a known allergy, or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components (including any of the constituents of the study vaccine)
* Participant has received respiratory syncytial virus (RSV) vaccine in a previous RSV vaccine study at any time prior to randomization

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (6):
- United States (6):
  - Optimal Research, Huntsville, Alabama
  - Optimal Research, San Diego, California
  - Optimal Research, Melbourne, Florida
  - Optimal Research, Peoria, Illinois
  - Optimal Research, Rockville, Maryland
  - Optimal Research, Austin, Texas

REFERENCES:
- [Derived] Comeaux CA, Bart S, Bastian AR, Klyashtornyy V, De Paepe E, Omoruyi E, van der Fits L, van Heesbeen R, Heijnen E, Callendret B, Sadoff J. Safety, Immunogenicity, and Regimen Selection of Ad26.RSV.preF-Based Vaccine Combinations: A Randomized, Double-blind, Placebo-Controlled, Phase 1/2a Study. J Infect Dis. 2024 Jan 12;229(1):19-29. doi: 10.1093/infdis/jiad220. PMID 37433021

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Pooled Placebo: Participants received a single intramuscular (IM) injection of placebo on Day 1, Day 57 and at Month 12 in Groups 1, 3, and 6. In Group 8, participants received single IM injection of placebo in each arm on Day 1 and at Month 12 and then a single placebo IM injection in one arm alone on Day 57.
- Cohort 1: RSV preF Protein 50 mcg: Participants received a single IM injection of respiratory syncytial virus (RSV) pre-fusion (preF) protein 50 micrograms (mcg) on Day 1, Day 57 and at Month 12 in Group 2 of Cohort 1.
- Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture): Participants received a single IM injection of a mixture of adenovirus serotype 26 RSV preF (Ad26.RSV.preF) 5*10^10 viral particles (vp) plus RSV preF protein 50 mcg on Day 1, Day 57 and at Month 12 in Group 4 of Cohort 1.
- Cohort 1: RSV preF Protein 150 mcg: Participants received a single IM injection of RSV preF protein 150 mcg on Day 1, Day 57 and at Month 12 in Group 5 of Cohort 1.
- Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture): Participants received a single IM injection of a mixture of Ad26.RSV.preF 5*10^10 vp plus RSV preF protein 150 mcg on Day 1, Day 57 and at Month 12 in Group 7 of Cohort 1.
- Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg in one arms on Day 1, Day 57, and at Month 12 and placebo IM injection in another arm on Day 1 and at Month 12 in Group 9 of Cohort 1.
- Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone: Participants received a single IM injection of Ad26.RSV.preF 1*10^11 vp in one arm and RSV preF protein 150 mcg IM injection in another arm on Day 1 and at Month 12, and placebo IM injection alone on Day 57 in Group 10 of Cohort 1.
- Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone: Participants received a single IM injection of Ad26.RSV.preF 1*10^11 vp in one arm and placebo in another arm on Day 1, followed by single IM injection of placebo alone on Day 57 in Group 11 of Cohort 2.
- Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 5*10^10 vp plus RSV preF protein 50 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo alone on Day 57 in Group 12 of Cohort 2.
- Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 50 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo alone on Day 57 in Group 13 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo alone on Day 57 in Group 14 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 5*10^10 vp plus RSV preF protein 150 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo alone on Day 57 in Group 15 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone: Participants received a single IM injection of Ad26.RSV.preF 1*10^11 vp in one arm and RSV preF protein 150 mcg in another arm on Day 1, followed by a single IM injection of placebo alone on Day 57 in Group 16 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg in one arm on Day 1 and Day 57 and a single IM injection of placebo in another arm on Day 1 in Group 17 of Cohort 2.
- Cohort 2: Pooled Placebo: Participants received two IM injections of placebo, one on each arm, on Day 1 and a single IM injection of placebo on Day 57 in Group 18 of Cohort 2.
- Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture): Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg (Cohort 2 selected regimen) on Day 1, Month 12, and Month 24 in Group 19 of Cohort 3.
- Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg (Cohort 2 selected regimen) on Day 1 and Month 24 and a placebo alone on Month 12 in Group 20 of Cohort 3.
- Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen: Participants received a single IM injection of Cohort 2 selected regimen and a placebo on Day 1, Month 12, and Month 24 in Group 21 of Cohort 3.
Period: Overall Study
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Started | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 24 | 42 | 42 | 42 | 43 | 36 | 36 | 24 | 135 | 136 | 45
Randomized and Vaccinated (Full Analysis Set) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24 | 135 | 136 | 44
Completed | 14 | 7 | 8 | 7 | 8 | 6 | 8 | 16 | 37 | 34 | 27 | 17 | 29 | 32 | 20 | 76 | 75 | 24
Not Completed | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 8 | 5 | 8 | 15 | 26 | 7 | 4 | 4 | 59 | 61 | 21
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 4 | 9 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 2 | 12 | 23 | 5 | 3 | 3 | 43 | 44 | 18
Not completed — Sponsor's Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Initiated Prohibited Medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4 | 1 | 0
Not completed — Randomized but not vaccinated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were randomized and received at least one dose of vaccine (active or placebo), regardless of the occurrence of protocol deviations or the type of vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen | Total
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24 | 135 | 136 | 44 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.22) | 67 (6.05) | 67.4 (6.21) | 69.4 (6.23) | 67.3 (3.88) | 64.5 (3.78) | 66.1 (6.17) | 68.5 (6.29) | 69 (6.9) | 68.5 (6.96) | 67.5 (5.71) | 71 (7.58) | 69 (6.49) | 66.5 (5.03) | 69 (7.08) | 67.9 (6.43) | 68.4 (6.25) | 69.3 (6.12) | 68.3 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 4 | 5 | 5 | 5 | 4 | 13 | 24 | 27 | 28 | 27 | 20 | 28 | 13 | 83 | 78 | 24 | 400
  Male | 8 | 4 | 4 | 3 | 3 | 3 | 4 | 11 | 18 | 15 | 14 | 15 | 16 | 8 | 11 | 52 | 58 | 20 | 267
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 6 | 3 | 4 | 1 | 4 | 3 | 9 | 1 | 38
  Not Hispanic or Latino | 16 | 8 | 7 | 8 | 8 | 7 | 8 | 22 | 41 | 39 | 36 | 39 | 32 | 35 | 20 | 132 | 127 | 43 | 628
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4
  Asian | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 0 | 1 | 0 | 4 | 4 | 4 | 3 | 0 | 2 | 3 | 2 | 5 | 3 | 11 | 16 | 0 | 62
  White | 12 | 4 | 8 | 7 | 7 | 3 | 4 | 20 | 37 | 40 | 38 | 36 | 34 | 31 | 21 | 121 | 117 | 41 | 581
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 16 | 8 | 8 | 8 | 8 | 8 | 8 | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24 | 135 | 136 | 44 | 667

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important. The outcome measure was planned to be analyzed for specified arms only.
Time Frame: From Day 1 up to Day 730
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
Participants | 3 | 0 | 0 | 2 | 3 | 0 | 0

2. Primary Outcome: Cohort 2 (Groups 11-13 and 16-18): Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From Day 1 up to Day 730
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 24 | 42 | 42 | 36 | 36 | 24
Participants | 0 | 5 | 5 | 7 | 3 | 4

3. Primary Outcome: Cohort 2 (Groups 14-15): Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From Day 1 up to Day 1095
Population: The FAS included all participants who were randomized and received at least one dose of vaccine (active or placebo), regardless of the occurrence of protocol deviations or the type of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone
Number analyzed (Participants) | 42 | 42
Participants | 4 | 5

4. Primary Outcome: Cohort 3: Number of Participants With Serious Adverse Events (SAEs)
Description: as for outcome 1
Time Frame: From Day 1 up to Day 1095
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 135 | 136 | 44
Participants | 14 | 16 | 3

5. Primary Outcome: Cohort 1: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 1
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 1 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local (injection site) AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post-vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 1 on Day 1 (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Pooled Placebo: Participants received a single intramuscular (IM) injection of placebo on Day 1, Day 57 and at Month 12 in Groups 1, 3, and 6 of Cohort 1. In Group 8, participants received single IM injection of placebo in each arm on Day 1 and at Month 12 and then a single placebo IM injection in one arm alone on Day 57.
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
Participants
  Solicited Local AEs | 3 | 2 | 4 | 0 | 5 | 6 | 6
  Solicited Systemic AEs | 4 | 0 | 4 | 1 | 4 | 5 | 5

6. Primary Outcome: Cohort 1: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 2
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 2 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants will be specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 2 on Day 57 (Day 64)
Population: The FAS included all participants who were randomized and received at least one dose of vaccine (active or placebo), regardless of the occurrence of protocol deviations or the type of vaccine. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 15 | 6 | 8 | 8 | 8 | 8 | 8
Participants
  Solicited Local AEs | 5 | 1 | 3 | 2 | 3 | 7 | 0
  Solicited Systemic AEs | 5 | 0 | 1 | 3 | 4 | 3 | 1

7. Primary Outcome: Cohort 1: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 3
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 3 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 3 on Day 365 (Day 372)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 11 | 8 | 8 | 7 | 7 | 6 | 8
Participants
  Solicited Local AEs | 1 | 0 | 3 | 2 | 4 | 5 | 6
  Solicited Systemic AEs | 2 | 1 | 0 | 2 | 5 | 0 | 3

8. Primary Outcome: Cohort 2: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 1
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 1 in Cohort 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 1 on Day 1 (Day 8)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 5*10^10 vp plus RSV preF protein 50 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo on Day 57 in Group 12 of Cohort 2.
- Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 50 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo on Day 57 in Group 13 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo on Day 57 in Group 14 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone: Participants received a single IM injection of a mixture of Ad26.RSV.preF 5*10^10 vp plus RSV preF protein 150 mcg in one arm and single IM injection of placebo in another arm on Day 1, followed by a single IM injection of placebo on Day 57 in Group 15 of Cohort 2.
- Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone: Participants received a single IM injection of Ad26.RSV.preF 1*10^11 vp in one arm and RSV preF protein 150 mcg in another arm on Day 1, followed by a single IM injection of placebo on Day 57 in Group 16 of Cohort 2.
- Cohort 2: Pooled Placebo: Participants received two IM injections of placebo in separate arms on Day 1 and single IM injection on Day 57 in Group 18 of Cohort 2.
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24
Participants
  Solicited Local AEs | 14 | 24 | 26 | 29 | 25 | 20 | 22 | 5
  Solicited Systemic AEs | 11 | 23 | 20 | 22 | 21 | 20 | 20 | 11

9. Primary Outcome: Cohort 2: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 2
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 2 in Cohort 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 2 on Day 57 (Day 64)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 23 | 40 | 38 | 42 | 42 | 33 | 35 | 23
Participants
  Solicited Local AEs | 1 | 0 | 3 | 3 | 3 | 2 | 23 | 2
  Solicited Systemic AEs | 3 | 9 | 8 | 7 | 5 | 5 | 13 | 6

10. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 1
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 1 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 1 on Day 1 (Day 8)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo: Participants received a single IM injection of a mixture of Ad26.RSV.preF 1*10^11 vp plus RSV preF protein 150 mcg (Cohort 2 selected regimen) on Day 1 and Month 24, followed by matching placebo alone on Month 12 in Group 20 of Cohort 3.
- Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen: Participants received a single IM injection of Cohort 2 selected regimen matching placebo on Day 1, Month 12, and Month 24 in Group 21 of Cohort 3.
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 134 | 136 | 44
Participants
  Solicited Local AEs | 95 | 94 | 9
  Solicited Systemic AEs | 95 | 88 | 12

11. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 2
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 2 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 2 on Day 365 (Day 372)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 112 | 114 | 38
Participants
  Solicited Local AEs | 74 | 23 | 6
  Solicited Systemic AEs | 56 | 38 | 10

12. Primary Outcome: Cohort 3: Number of Participants With Solicited Local (Injection Site) and Systemic AEs at 7 Days Post-vaccination 3
Description: Number of participants with solicited local and systemic AEs at 7 days post-vaccination 3 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, are used to assess the reactogenicity of the study vaccine and are pre-defined local (injection site). Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: 7 days post-vaccination 3 on Day 730 (Day 737)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 73 | 73 | 25
Participants
  Solicited Local AEs | 42 | 48 | 4
  Solicited Systemic AEs | 32 | 46 | 6

13. Primary Outcome: Cohort 1: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 1
Description: Number of participants with unsolicited AEs post-vaccination 1 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 1 on Day 1 (Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
Participants | 2 | 5 | 0 | 1 | 3 | 4 | 3

14. Primary Outcome: Cohort 1: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 2
Description: Number of participants with unsolicited AEs post-vaccination 2 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 2 on Day 57 (Day 85)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 15 | 6 | 8 | 8 | 8 | 8 | 8
Participants | 2 | 1 | 2 | 0 | 2 | 4 | 0

15. Primary Outcome: Cohort 1: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 3
Description: Number of participants with unsolicited AEs post-vaccination 3 in Cohort 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 3 on Day 365 (Day 393)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 11 | 8 | 8 | 7 | 7 | 6 | 8
Participants | 1 | 0 | 0 | 1 | 0 | 1 | 1

16. Primary Outcome: Cohort 2: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 1
Description: Number of participants with unsolicited AEs post-vaccination 1 in Cohort 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 1 on Day 1 (Day 29)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24
Participants | 8 | 11 | 10 | 12 | 8 | 10 | 12 | 3

17. Primary Outcome: Cohort 2: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 2
Description: Number of participants with unsolicited AEs post-vaccination 2 in Cohort 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 2 on Day 57 (Day 85)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 23 | 40 | 38 | 42 | 42 | 33 | 35 | 23
Participants | 6 | 5 | 5 | 6 | 2 | 3 | 5 | 8

18. Primary Outcome: Cohort 3: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 1
Description: Number of participants with unsolicited AEs post-vaccination 1 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 1 on Day 1 (Day 29)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 134 | 136 | 44
Participants | 32 | 23 | 7

19. Primary Outcome: Cohort 3: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 2
Description: Number of participants with unsolicited AEs post-vaccination 2 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 2 on Day 365 (Day 393)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 112 | 114 | 38
Participants | 9 | 10 | 4

20. Primary Outcome: Cohort 3: Number of Participants With Unsolicited AEs at 28 Days Post-vaccination 3
Description: Number of participants with unsolicited AEs post-vaccination 3 in Cohort 3 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs are all AEs for which the participant is not specifically questioned in the participant diary.
Time Frame: 28 days post-vaccination 3 on Day 730 (Day 758)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 73 | 73 | 25
Participants | 8 | 8 | 2

21. Primary Outcome: Cohort 2 (Group 11 to 15): Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers on Day 29
Description: RSV A2 Strain neutralization antibody titers on Day 29 was reported. Geometric mean titers (GMTs) of RSV A2 neutralizing antibodies were measured using the neutralization assay. The outcome measure was planned to be analyzed for specified arms only.
Time Frame: Day 29
Population: The per-protocol RSV immunogenicity (PPI) set included all participants who were randomized and received the complete first dose and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone
Number analyzed (Participants) | 22 | 40 | 42 | 42 | 42
Titers | 1642 [1165 to 2312] | 2869 [1964 to 4193] | 4813 [3642 to 6361] | 5189 [3730 to 7219] | 4855 [3865 to 6099]

22. Secondary Outcome: Cohort 1: RSV A2 Strain Neutralization Antibody Titers at Specified Timepoints
Description: RSV A2 strain neutralization antibody titers at specified timepoints in Cohort 1 was reported. The GMTs of RSV A2 neutralizing antibodies were measured using the neutralization assay.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, and 547
Population: PPI set included all participants who were randomized and received the complete first dose and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
Titers
  Day 1 | 553 [369 to 831] | 600 [301 to 1196] | 917 [474 to 1773] | 434 [301 to 625] | 457 [291 to 718] | 577 [364 to 915] | 522 [252 to 1082]
  Day 15: number analyzed (Participants) | 15 | 8 | 8 | 7 | 8 | 8 | 7
  Day 15 | 197 [103 to 378] | 4850 [2464 to 9547] | 823 [419 to 1620] | 644 [106 to 3919] | 1152 [640 to 2073] | 4404 [2122 to 9139] | 7782 [3715 to 16302]
  Day 29 | 412 [268 to 632] | 3326 [1643 to 6732] | 5716 [2862 to 11416] | 4311 [1856 to 10016] | 5933 [3603 to 9770] | 2399 [1075 to 5352] | 3678 [1724 to 7848]
  Day 57: number analyzed (Participants) | 16 | 6 | 8 | 7 | 8 | 8 | 8
  Day 57 | 431 [288 to 646] | 3441 [1634 to 7245] | 5105 [2239 to 11639] | 3382 [1352 to 8460] | 5276 [2798 to 9947] | 3382 [1697 to 6738] | 3980 [1990 to 7964]
  Day 85: number analyzed (Participants) | 15 | 6 | 7 | 8 | 8 | 8 | 7
  Day 85 | 536 [348 to 827] | 4142 [2147 to 7991] | 4865 [1787 to 13248] | 4574 [2506 to 8346] | 4582 [2203 to 9531] | 4667 [2660 to 8189] | 3905 [1414 to 10788]
  Day 183: number analyzed (Participants) | 16 | 6 | 7 | 8 | 8 | 7 | 8
  Day 183 | 529 [324 to 864] | 2473 [882 to 6934] | 3889 [1691 to 8943] | 2444 [1186 to 5035] | 3438 [1505 to 7857] | 2759 [1388 to 5483] | 2073 [798 to 5389]
  Day 365: number analyzed (Participants) | 12 | 6 | 7 | 6 | 7 | 6 | 8
  Day 365 | 502 [350 to 719] | 595 [60 to 5857] | 2628 [889 to 7770] | 1395 [997 to 1952] | 2531 [1303 to 4915] | 2039 [1148 to 3621] | 1665 [714 to 3884]
  Day 393: number analyzed (Participants) | 8 | 5 | 4 | 3 | 4 | 5 | 6
  Day 393 | 442 [313 to 623] | 2548 [1135 to 5721] | 11814 [1048 to 133124] | 3468 [492 to 24453] | 3103 [1914 to 5030] | 2994 [1577 to 5682] | 3081 [1252 to 7581]
  Day 547: number analyzed (Participants) | 8 | 6 | 4 | 4 | 4 | 6 | 7
  Day 547 | 637 [327 to 1242] | 2149 [1119 to 4129] | 4613 [502 to 42401] | 2286 [865 to 6039] | 2359 [1077 to 5167] | 4080 [2732 to 6094] | 3548 [1599 to 7872]

23. Secondary Outcome: Cohort 3: RSV A2 Strain Neutralization Antibody Titers at Specified Timepoints
Description: RSV A2 strain neutralization antibody titers at specified timepoints in Cohort 3 was reported. The GMTs of RSV A2 neutralizing antibodies were measured using the neutralization assay.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, 547, 730, 744, 758
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 135 | 135 | 44
Titers
  Day 1 | 546 [487 to 612] | 552 [490 to 622] | 582 [460 to 738]
  Day 15: number analyzed (Participants) | 123 | 123 | 42
  Day 15 | 6739 [5875 to 7730] | 4982 [4375 to 5673] | 525 [379 to 727]
  Day 29: number analyzed (Participants) | 129 | 130 | 43
  Day 29 | 5808 [4981 to 6771] | 4338 [3767 to 4996] | 489 [394 to 607]
  Day 57: number analyzed (Participants) | 125 | 126 | 43
  Day 57 | 4412 [3657 to 5322] | 3891 [3314 to 4568] | 563 [448 to 707]
  Day 85: number analyzed (Participants) | 117 | 122 | 39
  Day 85 | 3765 [3220 to 4402] | 3252 [2829 to 3739] | 514 [399 to 661]
  Day 183: number analyzed (Participants) | 126 | 124 | 43
  Day 183 | 3220 [2787 to 3721] | 2829 [2482 to 3225] | 673 [533 to 849]
  Day 365: number analyzed (Participants) | 116 | 117 | 40
  Day 365 | 2021 [1706 to 2395] | 1895 [1641 to 2189] | 545 [413 to 720]
  Day 393: number analyzed (Participants) | 100 | 100 | 40
  Day 393 | 2856 [2453 to 3325] | 1741 [1487 to 2038] | 585 [453 to 755]
  Day 547: number analyzed (Participants) | 89 | 94 | 33
  Day 547 | 1743 [1484 to 2046] | 1364 [1160 to 1602] | 469 [353 to 622]
  Day 730: number analyzed (Participants) | 86 | 86 | 30
  Day 730 | 1051 [866 to 1277] | 841 [710 to 997] | 314 [242 to 407]
  Day 744: number analyzed (Participants) | 66 | 63 | 25
  Day 744 | 2116 [1790 to 2500] | 2473 [2004 to 3051] | 393 [280 to 552]
  Day 758: number analyzed (Participants) | 67 | 67 | 24
  Day 758 | 2201 [1852 to 2616] | 2315 [1783 to 3005] | 416 [293 to 589]

24. Secondary Outcome: Cohort 2 (Group 16): RSV A2 Strain Neutralization Antibody Titers on Day 29
Description: RSV A2 strain neutralization antibody titers on Day 29 in Group 16 of Cohort 2 was reported. The GMTs of RSV A2 neutralizing antibodies were measured using the neutralization assay. The outcome measure was planned to be reported for specified arms only.
Time Frame: Day 29
Population: PPI set included all participants who were randomized and received the complete first dose and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 34
Titers | 6053 [4770 to 7682]

25. Secondary Outcome: Cohort 2 (Group 17): RSV A2 Strain Neutralization Antibody Titers on Day 85
Description: RSV A2 strain neutralization antibody titers on Day 85 in Group 17 of Cohort 2 was reported. The GMTs of RSV A2 neutralizing antibodies were measured using the neutralization assay. The outcome measure was planned to be reported for specified arms only.
Time Frame: Day 85
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo
Number analyzed (Participants) | 34
Titers | 4616 [3395 to 6276]

26. Secondary Outcome: Cohort 1: Pre-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at Specified Timepoints
Description: GMT (ELISA units per liter [EU/L]) of RSV F-protein in pre-fusion form as assessed by ELISA at specified timepoints as assessed by ELISA at specified timepoints in Cohort 1 were reported.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, and 547
Population: PPI set included all participants who were randomized and received the complete first dose and for whom immunogenicity data were available. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
EU/L
  Day 1 | 245 [172 to 349] | 263 [100 to 695] | 360 [206 to 627] | 215 [152 to 306] | 274 [158 to 474] | 301 [174 to 521] | 242 [122 to 479]
  Day 15: number analyzed (Participants) | 15 | 8 | 8 | 7 | 8 | 8 | 7
  Day 15 | 261 [171 to 398] | 2144 [1026 to 4480] | 6121 [3251 to 11528] | 4315 [1277 to 14578] | 6268 [4664 to 8424] | 3507 [1854 to 6636] | 3396 [1286 to 8971]
  Day 29 | 219 [150 to 319] | 1697 [886 to 3252] | 4132 [2515 to 6789] | 3352 [1424 to 7889] | 3575 [2955 to 4324] | 2396 [1252 to 4583] | 2257 [1238 to 4115]
  Day 57: number analyzed (Participants) | 16 | 6 | 8 | 7 | 8 | 8 | 8
  Day 57 | 246 [166 to 363] | 1694 [840 to 3417] | 4715 [2526 to 8801] | 3450 [1223 to 9733] | 3469 [2218 to 5427] | 2339 [1253 to 4366] | 2145 [922 to 4986]
  Day 85: number analyzed (Participants) | 15 | 6 | 7 | 8 | 8 | 8 | 7
  Day 85 | 268 [176 to 408] | 2048 [750 to 5592] | 3768 [1843 to 7705] | 3996 [1727 to 9247] | 3215 [1998 to 5173] | 2672 [1822 to 3918] | 1688 [733 to 3887]
  Day 183: number analyzed (Participants) | 16 | 6 | 7 | 8 | 8 | 7 | 8
  Day 183 | 281 [172 to 460] | 1045 [379 to 2878] | 2105 [1265 to 3502] | 1715 [1023 to 2876] | 1415 [803 to 2493] | 1654 [998 to 2740] | 1095 [512 to 2332]
  Day 365: number analyzed (Participants) | 12 | 6 | 7 | 6 | 7 | 6 | 8
  Day 365 | 271 [183 to 402] | 365 [38 to 3500] | 1669 [997 to 2792] | 993 [571 to 1727] | 1192 [679 to 2093] | 1415 [836 to 2394] | 928 [444 to 1939]
  Day 393: number analyzed (Participants) | 8 | 5 | 4 | 3 | 4 | 5 | 6
  Day 393 | 333 [157 to 705] | 1259 [606 to 2617] | 3523 [2326 to 5337] | 2856 [476 to 17148] | 2796 [1425 to 5486] | 2970 [1790 to 4929] | 1952 [940 to 4050]
  Day 547: number analyzed (Participants) | 8 | 6 | 4 | 4 | 4 | 6 | 7
  Day 547 | 304 [160 to 579] | 952 [434 to 2086] | 2486 [839 to 7364] | 1813 [550 to 5975] | 1304 [1075 to 1581] | 2241 [1463 to 3433] | 1879 [1041 to 3391]

27. Secondary Outcome: Cohort 2: Pre-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at Specified Timepoints
Description: GMT (ELISA units per liter [EU/L]) of RSV F-protein in pre-fusion form as assessed by ELISA at specified timepoints as assessed by ELISA at specified timepoints in Cohort 2 were reported.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, and 547
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24
EU/L
  Day 1 | 436 [321 to 591] | 354 [278 to 452] | 278 [227 to 342] | 274 [206 to 365] | 318 [264 to 382] | 314 [239 to 413] | 326 [256 to 416] | 229 [172 to 304]
  Day 15: number analyzed (Participants) | 23 | 41 | 42 | 42 | 42 | 35 | 36 | 24
  Day 15 | 1239 [970 to 1581] | 3860 [3151 to 4728] | 3363 [2662 to 4250] | 6055 [4576 to 8012] | 5375 [4225 to 6838] | 4925 [3569 to 6796] | 5215 [3984 to 6827] | 217 [160 to 297]
  Day 29: number analyzed (Participants) | 22 | 40 | 42 | 42 | 42 | 34 | 36 | 24
  Day 29 | 912 [712 to 1167] | 2796 [2335 to 3348] | 2435 [1995 to 2973] | 3880 [3044 to 4946] | 3610 [2926 to 4454] | 3318 [2545 to 4324] | 3684 [2884 to 4706] | 234 [169 to 324]
  Day 57: number analyzed (Participants) | 23 | 39 | 40 | 41 | 42 | 30 | 36 | 23
  Day 57 | 1052 [826 to 1342] | 2397 [2016 to 2851] | 2150 [1736 to 2664] | 2977 [2429 to 3648] | 2853 [2397 to 3394] | 2521 [1981 to 3209] | 2903 [2330 to 3618] | 290 [208 to 403]
  Day 85: number analyzed (Participants) | 23 | 39 | 42 | 42 | 41 | 29 | 34 | 23
  Day 85 | 1028 [833 to 1270] | 2031 [1691 to 2441] | 1824 [1477 to 2252] | 2553 [2087 to 3122] | 2400 [2050 to 2811] | 1981 [1480 to 2651] | 2686 [2089 to 3455] | 289 [222 to 377]
  Day 183: number analyzed (Participants) | 23 | 38 | 42 | 41 | 41 | 29 | 34 | 23
  Day 183 | 699 [521 to 937] | 1086 [874 to 1349] | 1121 [902 to 1392] | 1369 [1104 to 1689] | 1320 [1108 to 1572] | 1083 [848 to 1383] | 1561 [1183 to 2060] | 251 [181 to 347]
  Day 365: number analyzed (Participants) | 19 | 38 | 39 | 40 | 38 | 28 | 33 | 20
  Day 365 | 612 [438 to 854] | 1027 [831 to 1268] | 868 [697 to 1081] | 990 [796 to 1230] | 1105 [934 to 1308] | 917 [725 to 1160] | 1230 [946 to 1601] | 204 [131 to 317]
  Day 547: number analyzed (Participants) | 16 | 34 | 33 | 35 | 31 | 27 | 29 | 19
  Day 547 | 554 [385 to 798] | 775 [618 to 973] | 779 [646 to 939] | 946 [772 to 1160] | 937 [797 to 1101] | 849 [651 to 1106] | 1072 [861 to 1333] | 264 [168 to 414]

28. Secondary Outcome: Cohort 1: Post-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at Specified Timepoints
Description: GMT (EU/L) of RSV F-protein in post-fusion form as assessed by ELISA at specified timepoints for Cohort 1 were reported.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, and 547
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
EU/L
  Day 1 | 222 [146 to 337] | 206 [71 to 593] | 316 [212 to 470] | 197 [134 to 290] | 210 [125 to 354] | 239 [115 to 494] | 159 [82 to 308]
  Day 15: number analyzed (Participants) | 15 | 8 | 8 | 7 | 8 | 8 | 8
  Day 15 | 194 [134 to 303] | 1208 [476 to 3069] | 4841 [2384 to 9831] | 2985 [622 to 14323] | 3032 [1699 to 5411] | 1739 [632 to 4790] | 973 [424 to 2233]
  Day 29 | 214 [143 to 318] | 986 [400 to 2432] | 3929 [2197 to 7028] | 2303 [891 to 5956] | 1698 [1225 to 2353] | 1499 [712 to 3156] | 1033 [607 to 1756]
  Day 57: number analyzed (Participants) | 16 | 6 | 8 | 7 | 8 | 8 | 8
  Day 57 | 217 [145 to 325] | 1164 [303 to 4473] | 3098 [1730 to 5550] | 964 [280 to 3321] | 864 [337 to 2216] | 866 [355 to 2113] | 693 [343 to 1400]
  Day 85: number analyzed (Participants) | 15 | 6 | 7 | 8 | 8 | 8 | 7
  Day 85 | 220 [141 to 342] | 1020 [285 to 3650] | 2122 [863 to 5214] | 1906 [824 to 4409] | 1332 [813 to 2184] | 1384 [760 to 2520] | 786 [369 to 1672]
  Day 183: number analyzed (Participants) | 16 | 6 | 7 | 8 | 8 | 7 | 8
  Day 183 | 254 [164 to 392] | 710 [189 to 2671] | 1827 [1059 to 3153] | 1163 [650 to 2079] | 844 [478 to 1492] | 857 [425 to 1726] | 547 [289 to 1037]
  Day 365: number analyzed (Participants) | 12 | 6 | 7 | 6 | 7 | 6 | 8
  Day 365 | 226 [148 to 347] | 225 [18 to 2874] | 1316 [834 to 2075] | 657 [288 to 1496] | 530 [280 to 1002] | 740 [401 to 1366] | 398 [196 to 807]
  Day 393: number analyzed (Participants) | 8 | 5 | 4 | 3 | 4 | 5 | 6
  Day 393 | 237 [106 to 530] | 874 [293 to 2609] | 2385 [1637 to 3476] | 1631 [206 to 12930] | 1408 [458 to 4333] | 1330 [497 to 3558] | 1140 [590 to 2199]
  Day 547: number analyzed (Participants) | 8 | 6 | 4 | 4 | 4 | 6 | 7
  Day 547 | 243 [114 to 516] | 607 [178 to 2071] | 1382 [1018 to 1877] | 863 [254 to 2936] | 723 [428 to 1221] | 1001 [550 to 1823] | 792 [447 to 1403]

29. Secondary Outcome: Cohort 2: Post-Fusion RSV Fusion Protein (F-protein) Geometric Mean Titers (GMTs) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at Specified Timepoints
Description: GMT (EU/L) of RSV F-protein in post-fusion form as assessed by ELISA at specified timepoints for Cohort 2 were reported.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, and 547
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo
Number analyzed (Participants) | 24 | 42 | 42 | 42 | 42 | 36 | 36 | 24
EU/L
  Day 1 | 270 [185 to 393] | 260 [204 to 332] | 228 [184 to 284] | 202 [146 to 278] | 237 [189 to 289] | 246 [188 to 323] | 234 [172 to 318] | 190 [135 to 267]
  Day 15: number analyzed (Participants) | 23 | 41 | 42 | 42 | 42 | 35 | 36 | 24
  Day 15 | 679 [509 to 906] | 1785 [1415 to 2251] | 1555 [1185 to 2040] | 2524 [1764 to 3611] | 2617 [1921 to 3564] | 2159 [1545 to 3015] | 2365 [1640 to 3410] | 181 [130 to 254]
  Day 29: number analyzed (Participants) | 22 | 40 | 42 | 42 | 42 | 34 | 36 | 24
  Day 29 | 612 [467 to 802] | 1542 [1233 to 1929] | 1233 [856 to 1775] | 2195 [1607 to 2999] | 2203 [1655 to 2933] | 1863 [1419 to 2444] | 1994 [1436 to 2769] | 219 [145 to 331]
  Day 57: number analyzed (Participants) | 23 | 39 | 40 | 41 | 42 | 30 | 36 | 23
  Day 57 | 634 [479 to 863] | 1403 [1162 to 1693] | 1239 [960 to 1598] | 1754 [1318 to 2333] | 1740 [1339 to 2262] | 1506 [1178 to 1929] | 1661 [1212 to 2277] | 257 [177 to 372]
  Day 85: number analyzed (Participants) | 23 | 39 | 42 | 42 | 41 | 29 | 34 | 23
  Day 85 | 513 [339 to 775] | 1144 [937 to 1398] | 1050 [825 to 1337] | 1397 [1061 to 1839] | 1400 [1064 to 1834] | 1088 [817 to 1450] | 1504 [1096 to 2065] | 241 [171 to 340]
  Day 183: number analyzed (Participants) | 23 | 38 | 42 | 41 | 41 | 29 | 34 | 23
  Day 183 | 455 [324 to 639] | 735 [583 to 926] | 727 [581 to 909] | 896 [667 to 1130] | 908 [716 to 1151] | 709 [565 to 889] | 924 [658 to 1297] | 232 [167 to 323]
  Day 365: number analyzed (Participants) | 19 | 38 | 39 | 40 | 38 | 28 | 33 | 20
  Day 365 | 409 [261 to 642] | 666 [537 to 825] | 605 [478 to 765] | 652 [501 to 847] | 785 [607 to 1015] | 660 [521 to 836] | 755 [547 to 1041] | 166 [97 to 281]
  Day 547: number analyzed (Participants) | 16 | 34 | 33 | 35 | 31 | 27 | 29 | 19
  Day 547 | 381 [234 to 621] | 507 [394 to 652] | 556 [445 to 693] | 640 [477 to 859] | 741 [562 to 977] | 570 [449 to 723] | 720 [543 to 956] | 222 [141 to 349]

30. Secondary Outcome: Cohort 1: Breadth of Interferon-gamma (IFN-gamma) T-Cells Responses Against RSV Analyzed by Enzyme-linked Immunospot (ELISpot) Assay at Specified Timepoints
Description: Breadth of IFN-gamma T-Cells responses against RSV analyzed by ELISpot assay at specified timepoints for Cohort 1 were reported. The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. The unit was Spot forming units (SFU)/10^6 peripheral blood mononuclear cells (PBMCs).
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, and 547
Population: as for outcome 26
Measure: Median (Full Range); unit: SFU/10^6 PBMCs
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 16 | 8 | 8 | 8 | 8 | 8 | 8
SFU/10^6 PBMCs
  Day 1: number analyzed (Participants) | 16 | 7 | 8 | 8 | 8 | 8 | 8
  Day 1 | 48 [6 to 254] | 39 [13 to 103] | 16 [5 to 121] | 26 [2 to 91] | 71 [12 to 182] | 34 [1 to 57] | 56 [16 to 175]
  Day 15: number analyzed (Participants) | 15 | 8 | 8 | 7 | 8 | 8 | 7
  Day 15 | 57 [10 to 286] | 341 [79 to 562] | 432 [102 to 1004] | 316 [177 to 876] | 390 [142 to 531] | 399 [158 to 631] | 480 [53 to 2696]
  Day 29: number analyzed (Participants) | 16 | 7 | 7 | 8 | 6 | 8 | 8
  Day 29 | 46 [1 to 193] | 211 [123 to 1190] | 183 [124 to 825] | 153 [20 to 380] | 271 [207 to 368] | 271 [110 to 397] | 416 [219 to 1910]
  Day 57: number analyzed (Participants) | 16 | 6 | 8 | 6 | 7 | 8 | 8
  Day 57 | 42 [8 to 225] | 78 [45 to 114] | 180 [32 to 491] | 130 [41 to 343] | 244 [121 to 461] | 167 [14 to 290] | 315 [143 to 2635]
  Day 85: number analyzed (Participants) | 15 | 5 | 6 | 8 | 7 | 8 | 6
  Day 85 | 52 [1 to 323] | 199 [169 to 482] | 398 [137 to 622] | 293 [131 to 590] | 556 [355 to 1229] | 432 [158 to 663] | 274 [181 to 3123]
  Day 183: number analyzed (Participants) | 16 | 6 | 7 | 8 | 8 | 7 | 5
  Day 183 | 56 [1 to 629] | 105 [33 to 386] | 281 [148 to 599] | 172 [74 to 271] | 301 [115 to 531] | 305 [144 to 472] | 215 [62 to 3022]
  Day 365: number analyzed (Participants) | 12 | 6 | 6 | 6 | 6 | 6 | 7
  Day 365 | 61 [21 to 312] | 152 [54 to 309] | 270 [171 to 582] | 158 [107 to 442] | 297 [128 to 531] | 231 [136 to 594] | 249 [117 to 2021]
  Day 393: number analyzed (Participants) | 8 | 5 | 4 | 2 | 3 | 4 | 6
  Day 393 | 54 [3 to 411] | 159 [93 to 584] | 492 [321 to 811] | 472 [211 to 733] | 720 [614 to 1000] | 400 [25 to 726] | 443 [248 to 2362]
  Day 547: number analyzed (Participants) | 8 | 6 | 4 | 4 | 4 | 6 | 7
  Day 547 | 42 [11 to 737] | 199 [67 to 306] | 262 [197 to 397] | 245 [107 to 308] | 374 [195 to 387] | 202 [85 to 505] | 258 [96 to 2443]

31. Secondary Outcome: Cohort 3: Breadth of Interferon-gamma (IFN-gamma) T-Cells Responses Against RSV Analyzed by Enzyme-linked Immunospot (ELISpot) Assay at Specified Timepoints
Description: Breadth of IFN-gamma T-Cells responses against RSV analyzed by ELISpot assay at specified timepoints for Cohort 3 were reported. The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. The unit was SFU/10^6 PBMCs.
Time Frame: Days 1, 15, 29, 57, 85, 183, 365, 393, 730, 744, and 758
Population: as for outcome 22
Measure: Median (Full Range); unit: SFU/10^6 PBMCs
Arm/Group | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
Number analyzed (Participants) | 25 | 26 | 9
SFU/10^6 PBMCs
  Day 1: number analyzed (Participants) | 24 | 26 | 8
  Day 1 | 56 [5 to 612] | 73 [1 to 1030] | 39 [1 to 193]
  Day 15: number analyzed (Participants) | 25 | 25 | 9
  Day 15 | 515 [128 to 2308] | 566 [153 to 1563] | 17 [2 to 258]
  Day 29: number analyzed (Participants) | 25 | 25 | 9
  Day 29 | 348 [10 to 3179] | 457 [162 to 1089] | 46 [1 to 294]
  Day 57: number analyzed (Participants) | 23 | 20 | 8
  Day 57 | 371 [122 to 3614] | 424 [181 to 2910] | 41 [2 to 264]
  Day 85: number analyzed (Participants) | 23 | 22 | 8
  Day 85 | 301 [103 to 3770] | 327 [58 to 3187] | 18 [18 to 499]
  Day 183: number analyzed (Participants) | 24 | 22 | 8
  Day 183 | 218 [60 to 3710] | 227 [18 to 3186] | 32 [7 to 211]
  Day 365: number analyzed (Participants) | 23 | 21 | 9
  Day 365 | 152 [40 to 3261] | 233 [61 to 2896] | 44 [1 to 123]
  Day 393: number analyzed (Participants) | 20 | 20 | 9
  Day 393 | 364 [92 to 994] | 207 [41 to 2634] | 30 [2 to 211]
  Day 547: number analyzed (Participants) | 20 | 16 | 8
  Day 547 | 284 [94 to 6756] | 233 [37 to 2108] | 17 [1 to 166]
  Day 730: number analyzed (Participants) | 19 | 15 | 7
  Day 730 | 210 [103 to 5930] | 243 [41 to 1873] | 25 [14 to 64]
  Day 744: number analyzed (Participants) | 15 | 9 | 6
  Day 744 | 707 [213 to 5975] | 651 [390 to 1607] | 35 [6 to 65]
  Day 758: number analyzed (Participants) | 15 | 12 | 6
  Day 758 | 390 [84 to 5290] | 430 [264 to 2326] | 14 [1 to 25]

32. Secondary Outcome: Cohort 2 (Group 11-16): Breadth of IFN-gamma T-Cells Responses Against RSV Analyzed by ELISpot Assay on Day 29
Description: Breadth of IFN-gamma T-Cells responses against RSV analyzed by ELISpot Assay on Day 29 in Groups 11-16 of Cohort 2 was reported. The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. The outcome measure was planned to be analyzed for specified arms only.
Time Frame: Day 29
Population: The PPI set included all participants who were randomized and received the complete first dose and for whom immunogenicity data were available. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: SFU/10^6 PBMCs
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone
Number analyzed (Participants) | 18 | 33 | 33 | 35 | 34 | 31
SFU/10^6 PBMCs | 320 [203 to 592] | 354 [227 to 453] | 315 [192 to 497] | 290 [187 to 485] | 390 [251 to 586] | 298 [195 to 374]

33. Secondary Outcome: Cohort 2 (Group 17): Breadth of IFN-gamma T-Cells Responses Analyzed by ELISpot Assay on Day 85
Description: Breadth of IFN-gamma T-Cells responses analyzed by ELISpot assay on Day 85 in Group 17 of Cohort 2 was reported. The ELISPOT assay for F protein-specific gamma interferon-producing T cells was performed using RSV F peptides. The outcome measure was planned to be analyzed for specified arms only.
Time Frame: Day 85
Population: as for outcome 24
Measure: Median (Full Range); unit: SFU/10^6 PBMCs
Arm/Group | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo
Number analyzed (Participants) | 28
SFU/10^6 PBMCs | 495 [113 to 6855]

ADVERSE EVENTS:
Time Frame: From Day 1 up to 1095 days
Description: The full analysis set (FAS) included all participants who were randomized and received at least one dose of vaccine (active or placebo), regardless of the occurrence of protocol deviations or the type of vaccine.
Arm/Group | Cohort 1: Pooled Placebo | Cohort 1: RSV preF Protein 50 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) | Cohort 1: RSV preF Protein 150 mcg | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo | Cohort 2: Pooled Placebo | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/8 | 0/8 | 1/8 | 0/8 | 0/8 | 0/8 | 0/24 | 1/42 | 1/42 | 0/42 | 0/42 | 1/36 | 0/36 | 0/24 | 1/135 | 0/136 | 0/44
Serious Adverse Events (participants affected / at risk) | 3/16 | 0/8 | 0/8 | 2/8 | 3/8 | 0/8 | 0/8 | 0/24 | 5/42 | 5/42 | 4/42 | 5/42 | 7/36 | 3/36 | 4/24 | 14/135 | 16/136 | 3/44
Other Adverse Events (participants affected / at risk) | 5/16 | 5/8 | 2/8 | 2/8 | 4/8 | 6/8 | 4/8 | 12/24 | 14/42 | 14/42 | 15/42 | 10/42 | 10/36 | 15/36 | 10/24 | 25/135 | 27/136 | 13/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Pooled Placebo (N=16) | Cohort 1: RSV preF Protein 50 mcg (N=8) | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) (N=8) | Cohort 1: RSV preF Protein 150 mcg (N=8) | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) (N=8) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo (N=8) | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone (N=8) | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone (N=24) | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone (N=36) | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo (N=36) | Cohort 2: Pooled Placebo (N=24) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) (N=135) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo (N=136) | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen (N=44)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adverse Drug Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Portal Vein Thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis Infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colon Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malignant Palate Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Carotid Artery Occlusion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacunar Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Substance Abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Distributive Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemodynamic Instability (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Pooled Placebo (N=16) | Cohort 1: RSV preF Protein 50 mcg (N=8) | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 50 mcg (Mixture) (N=8) | Cohort 1: RSV preF Protein 150 mcg (N=8) | Cohort 1: Ad26.RSV.preF 5*10^10 vp + RSV preF Protein 150 mcg (Mixture) (N=8) | Cohort 1: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo (N=8) | Cohort 1: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone (N=8) | Cohort 2: Ad26.RSV.preF 1*10^11 vp With Placebo and Placebo Alone (N=24) | Cohort 2:Ad26.RSV.preF 5*10^10vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2:Ad26.RSV.preF 1*10^11vp + RSV preF Protein 50mcg(Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 1*10^11vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 5*10^10vp + RSV preF Protein 150mcg (Mixture) With Placebo and Placebo Alone (N=42) | Cohort 2: Ad26.RSV.preF 1*10^11 vp With RSV preF Protein 150 mcg and Placebo Alone (N=36) | Cohort 2: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) Alone and With Placebo (N=36) | Cohort 2: Pooled Placebo (N=24) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) (N=135) | Cohort 3: Ad26.RSV.preF 1*10^11 vp + RSV preF Protein 150 mcg (Mixture) and Placebo (N=136) | Cohort 3: Pooled Placebo of Cohort 2 Selected Regimen (N=44)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trichiasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukoplakia Oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary Gland Enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection Site Erosion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection Site Haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection Site Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to Arthropod Bite (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 8 | 4 | 5 | 1 | 3 | 5 | 5 | 3 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Tooth Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Animal Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Diastolic Increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Systolic Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic Keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous Cell Carcinoma of Head and Neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balance Disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Dizziness Postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Venous Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03502707/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/07/NCT03502707/SAP_001.pdf